CLINICAL TRIAL: NCT06676579
Title: A Multi-Center, Phase II, Open Label, Randomized Trial Evaluating the Efficacy and Safety of Complement 5a Receptor Antagonist Avacopan in Crescentic IgA Nephropathy
Brief Title: Avacopan in Crescentic Immunoglobulin A Nephropathy (IgAN)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fernando Fervenza, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-005668
Record Dates: First submitted 2024-10-29; First posted 2024-11-06 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: IgA Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — avacopan; Prednisone; Methylprednisolone; Pharmaceutical Preparations; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avacopan and Low Doses Glucocorticoid (Active Comparator): * Methylprednisolone 1g intravenous on day +1
  * Prednisone 0.2 mg/kg per day (maximum, 16 mg/day) for 2 months followed by dose tapering by 2 mg per day each month (total duration 6-9 months)
  * Avacopan 30 mg oral twice a day (1-0-1) for 12 months
  Interventions: Drug: Avacopan; Drug: Methylprednisolone (drug); Drug: Prednisolone
- High Doses Glucocorticoid (Active Comparator): * Methylprednisolone 1g intravenous on day +1
  * Prednisone 0.4 mg/kg per day (maximum, 32 mg/day) for 2 months followed by dose tapering by 4 mg per day each month (total duration 6-9 months)
  Interventions: Drug: Prednisone; Drug: Methylprednisolone (drug)

INTERVENTIONS:
Drug: Avacopan — Avacopan is a complement 5a receptor (C5aR) antagonist, orally active.
  Other Names: Tavneos
  Arms: Avacopan and Low Doses Glucocorticoid
Drug: Prednisone — 0.4 mg/kg per day (maximum, 32 mg/day) for 2 months followed by dose tapering by 4 mg per day each month (total duration 6-9 months
  Arms: High Doses Glucocorticoid
Drug: Methylprednisolone (drug) — Methylprednisolone 1g intravenous on day +1
Drug: Prednisolone — Prednisone 0.2 mg/kg per day (maximum, 16 mg/day) for 2 months followed by dose tapering by 2 mg per day each month (total duration 6-9 months)
  Arms: Avacopan and Low Doses Glucocorticoid

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Avacopan together with low-dose glucocorticoid in the treatment of patients with crescentic Imunoglobulin A Nephropathy (IgAN) and high risk of progression.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years
* Kidney biopsy showing crescentic IgA nephropathy within 6 months of enrolment (MEST-C-score =C1/C2).
* Quantified creatinine clearance >20 ml/min/1.73m2
* Quantified Proteinuria > 750 mg/24h based on a 24h urine collection while on maximum tolerated dose of RAS blockade
* Hematuria defined as >10 RBC/hpf or hemoglobinuria >1+
* Patients need to be in adequate supportive care (blood pressure <125/85mmHg, lifestyle advice, and maximum doses tolerable of RAS blockade) at least 4 weeks prior to enrollment
* Patients would receive dietary and lifestyle counseling prior enrollment: low protein (0.8-1.0 g/kg/day) diet, low sodium (2 grams/day) intake, indication for smoke cessation, during the 4 weeks run-in period
* Has signed an informed consent form prior to any study-related procedures
* Patients with documented use of RAS blockade and adequate blood pressure control (<125/85 mmHg) for ≥4 weeks, can be enrolled in the study and randomized without repeating a 4-week run-in period.

Exclusion Criteria

* Creatinine clearance <20 ml/min/1.73 m2
* Liver function tests > 2x upper limit of normal. (Serious cases of hepatotoxicity have been reported in patients with avacopan during first approval and ADVOCATE study (29) (30)
* Severe interstitial fibrosis and tubular atrophy (IFTA > 70% on renal biopsy)
* Active cancer or acute non-controlled infection (including HIV, HBV, HCV)
* Women who are pregnant or breastfeeding
* Immunosuppression treatment:
* Rituximab less than 12 months prior to enrollment
* MMF, CYC, or immunomodulatory agents within 3 months prior to enrollment
* AZA within 3 months prior to enrollment.
* Glucocorticoids >20 mg/day within 1 month prior to enrollment
* Secondary IgA nephropathy (associated with gastrointestinal diseases, infection, autoimmune, malignancy, respiratory tract, or skin)
* ANCA-associated vasculitis or other vasculitis diagnostic defined by ACR criteria/Chapel Hill Consensus conference
* Contraindication to use any of the protocol treatments (glucocorticoids, avacopan)
* Use of a strong/moderate CYP3A4 inducer
* Initiation of SGLT2 inhibitors is not allowed once patient has been enrolled in the study. Patients who have been on an SGLT2 inhibitor prior to enrollment on the study may continue on this therapy, at the same dose. No dose increase is allowed.
* Active, untreated and/or uncontrolled chronic liver disease (chronic active hepatitis B, untreated hepatitis C, uncontrolled autoimmune hepatitis, cirrhosis
* Unable to give written consent form
* As a safety measure patients who are pregnant or lactating will not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-03-02 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in proteinuria measured by results of protein total, 24-hour urine collection at baseline compared to collection at 12 months. | 12 months
  A response is based on the average of proteinuria quantified twice over a 2-weeks period at 12 months.

SECONDARY OUTCOMES:
Change in proteinuria >50% | 12 months
  This is based on the average of proteinuria quantified twice over a 2-weeks period at 12 months.
Change in eGFR (using 2021 CKD-EPI Formula) | 6 months, 12 months
  • Change in eGFR (using 2021 CKD-EPI Formula) at 6 and 12 months compared to baseline
Change in hematuria from Baseline to 12 month visit. | 12 months
  Hematuria is measured in the urinalysis done at baseline and 12-month visit.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fervenza, MD, Principal Investigator — Mayo Clinic, Rochester, MN; Nabeel Aslam, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No